CLINICAL TRIAL: NCT02699229
Title: Non-linear Multimodal Microendoscopy for Lung Cancer Pathology
Status: Withdrawn | Type: Observational
Why Stopped: no particpants enrolled
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-7485
Record Dates: First submitted 2015-12-02; First posted 2016-03-04 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Malignant: Tissue sample
- Benign: Tissue sample
- Normal: Tissue Sample

SUMMARY:
For this study the investigators are looking to do the following:

1. To characterize human lung lesions by nonlinear microscopy using ex vivo tissues.
2. To establish the first spectral/structural database for nonlinear optical microimaging of normal and abnormal lung tissue.

DETAILED DESCRIPTION:
For this study the investigators are looking to do the following:

1. To characterize human lung lesions by nonlinear microscopy using ex vivo tissues. In particular, to investigate collagen content and ultrastructure with SHG (second harmonic generation) microscopy, to characterize cell and nuclear morphology and lipid vesicle content with THG (third harmonic generation) and CARS (coherent anti-Stokes Raman scattering) microscopy and to conduct spectroscopic and lifetime characterization of MPF (multiphoton fluorescence) signals in cancerous, benign, and normal tissues.
2. To establish the first spectral/structural database for nonlinear optical microimaging of normal and abnormal lung tissue, from which to generate diagnostic algorithms, both to optimize the operating parameters of planned nonlinear endoscopic imaging and to serve as the basis for nonlinear optical histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients with confirmed or suspected lung cancer who require lobectomy as part of standard-of-care.

Exclusion Criteria:

* Patients deemed on clinical grounds not to be medically fit for a lobectomy
* Patients where there is a high clinical suspicion of lymphoma (to avoid mixing the data sets).
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Nonlinear optical microscopy for cancerous tissue detection in human lung lesions | Two years

SECONDARY OUTCOMES:
The first spectral/structural database for nonlinear optical micro-imaging of normal and abnormal lung tissue | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku, MD, PhD, Principal Investigator — University Health Network, Toronto